CLINICAL TRIAL: NCT02245204
Title: Phase I Studies of Chlorogenic Acid for Injection for Tolerance and Pharmacokinetic of Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan J.Z. Bio-chemical Science and Technology Development Co., Ltd (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYS-I-01
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Chlorogenic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chlorgenic acid, Treatment, powder (Experimental): Chlorogenic acid for injection(30mg/bottle) is white or off-white freeze-dried lump or powder,it can be easily dissolved in water, which solubility is 20%.
  Interventions: Drug: Chlorogenic acid

INTERVENTIONS:
Drug: Chlorogenic acid — Chlorogenic acid for injection is polyphenols, micromolecular and un-endogenous substance. It might play the role of cancer treatment via balancing tumor micro-environmental immune status according to the stability and rationality of immunodeficiency and endogenous immune material expression around the tumor. Chlorogenic acid for injection is made from chlorogenic acid (purity≥98%) which is extracted from folium cortex eucommiae.Chlorogenic acid and its preparations have not been reported as chemical drug and marketed around the world.

SUMMARY:
The purpose of this study:

Determining the Maximum Tolerated Dose (MTD), Dose-Limiting Toxicity (DLT), pharmacokinetics characteristic, and dosage regimen of phase II/III of Chlorogenic acid for injection in the advanced malignant tumor subjects;

DETAILED DESCRIPTION:
1. Investigate the tolerance of Chlorogenic acid for injection in human body, determine the Maximum Tolerated Dose (MTD) and Dose-Limiting Toxicity (DLT) of Chlorogenic acid for injection in the advanced malignant tumor subjects;
2. Determine the human pharmacokinetics characteristic of Chlorogenic acid for injection;
3. Preliminary observation the effectiveness and effective dose;
4. Provide the basis for the dosage regimen of phase II/III.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologic or/and FNAC confirmation of advanced cancer but without effective treatment or with treatment failure;
2. Between 18 and 65 years of age, KPS≥70;
3. According to RECIST 1.1,patients with at least one tumor lesion that can accurately be measured by CT or MRI in at least one dimension with longest diameter to be recorded as >2.0cm by general CT or >1.0cm by spiral CT;
4. Life expectancy of at least three (3) months at the enrollment;
5. Patients who have sufficient baseline organ function and whose laboratory data can meet the following criteria at the enrollment:

   * PLT count≥100×10~9/L,
   * WLB count≥4.0×10~9/L and ≤12×10~9/L,
   * Neutrophil granulocyte count≥2.0×10~9/L,
   * HGB count≥90g/L,
   * Total bilirubin <=1.5 times of ULN,
   * ALT/AST ≤2.5 times of ULN,
   * SCr≤1.5 times of ULN,
   * Normal ECG with LVEF (≥50%) measured by echocardiography;
6. Female patients with negative pregnant test, and male/female patients of reproductive age without pregnancy planning in the next 12 months;
7. Volunteered for the phase 1 trial and sign the informed consent without protest;

Exclusion Criteria:

1. Patients who have received large area radiotherapy （>30% marrow capacity）;
2. Patients who suffer from other serious complication, such as uncontrollable infection, myocardial infarction within the past 6 months at the enrollment , uncontrollable hypertension ,thromboembolism and etc.;
3. Symptomatic patients with brain metastases (except for the patients whose brain metastases is controlled to stable status after whole brain radiotherapy);
4. Patients who have received the therapy of chemotherapy within 4 weeks before enrollment;
5. Patients who have used nitrosoureas drug or mitomycin within 6 weeks or tyrosine kinase inhibitor within 2 weeks before enrollment;
6. Patients who have received therapy of major surgery within 6 weeks or biopsy surgery within 2 weeks before enrollment;
7. Patients who or have received radical radiotherapy within 6 weeks or local palliative radiotherapy within 2 weeks before enrollment;
8. Patients who experience grade 2 or more than grade 2 toxicity caused by the past therapies;
9. Patients who have history of drug abuse or alcoholism;
10. Patients who smoke over 5 cigarettes or equivalent tobacco per day;
11. Uncontrollable psychopaths;
12. Pregnant or breast-feeding women, or patients(male and female) who have pregnancy plan;
13. Patients who had received a therapy of another investigational drug within 4 weeks or patients who are still in another clinical trial at the enrollment;
14. Known active hepatitis B/hepatitis C, positive HIV/ syphilis antibody;
15. Patient who need long term treatment of cortical hormone or other immunosuppressive drugs such as visceral organ transplanters;
16. Allergic to the investigational drug;
17. Other patients judged ineligible for enrollment in the study by the investigator (sub-investigator).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Within the first 60 days after the first dose of chlorogenic acid

SECONDARY OUTCOMES:
Dose-Limiting Toxicity | Within the first 30 days after the first dose of chlorogenic acid
Maximum Tolerated Dose | Within the first 30 days after the first dose of chlorogenic acid
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of chlorogenic acid | Within the first 30 days after the first dose of chlorogenic acid
Improvement in cancer-related symptoms and quality of life | Within 1 year after the first dose of chlorogenic acid

OTHER OUTCOMES:
Changing in number of red blood cell and level of hemoglobin | within 1 year after the first dose of chlorogenic acid
Changing in the diameters of lymph node metastasis | Within 1 year after the first dose of chlorogenic acid
Changing in levels of tumor markers | Within 1 year after the first dose of chlorogenic acid

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Dr, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China